CLINICAL TRIAL: NCT06994585
Title: Comparing the Bowel Cleansing Efcacy of Picosulfate Sodium/ Citric Acid / Magnesium Oxide and Polyethylene Glycol: A Randomized Trial in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Drinklear study
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2023-12

CONDITIONS: Bowel Preparation
Keywords: Drinklear powder，Niflec Powder，Picosulfate Sodium/ Citric Acid / Magnesium Oxide， Polyethylene Glycol，Bowel Cleansing Efcacy，bowel preparation

STUDY DESIGN:
Intervention Model Description: Inclusion criteria include outpatient patients at our institution, aged 20 to 75 years, who are scheduled to undergo colonoscopy and are willing to participate in this research study. Exclusion criteria comprise patients with allergies to bowel preparation agents, those who fail to show up on the scheduled date, patients who refuse to participate, those unable to follow preparation instructions, individuals with intestinal perforation, gastric retention, gastrointestinal obstruction, or bowel obstruction, severe renal insufficiency (CrCl below 30 mL/min), pregnant individuals, toxic megacolon, and patients with colorectal cancer.
  Statistical Analysis Plan for this study: This is a non-inferiority study with a one-sided non-inferiority hypothesis. The non-inferiority margin is set at 0.1. The sample size for each group is 220, resulting in a total of 440 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drinklear (Experimental): sodium picosulfate/magnesium citrate
  Interventions: Drug: Drinklear
- Niflec (Experimental): Polyethylene Glycol
  Interventions: Drug: Niflec

INTERVENTIONS:
Drug: Drinklear — Our hospital invites outpatient patients aged 20 to 75 years who are scheduled to undergo colonoscopy and are willing to participate in this research study. After obtaining informed consent and signing the consent form, participants will be randomly assigned to receive either Polyethylene Glycol (Niflec Powder, China Chemical & Pharmaceutical Co., Ltd., Taiwan) or Picosulfate Sodium/Citric Acid/Magnesium Oxide (Drinklear Powder, China Chemical & Pharmaceutical Co., Ltd., Taiwan) as the bowel preparation for colonoscopy.
  Arms: Drinklear
Drug: Niflec — Our hospital invites outpatient patients aged 20 to 75 years who are scheduled to undergo colonoscopy and are willing to participate in this research study. After obtaining informed consent and signing the consent form, participants will be randomly assigned to receive either Polyethylene Glycol (Niflec Powder, China Chemical & Pharmaceutical Co., Ltd., Taiwan) or Picosulfate Sodium/Citric Acid/Magnesium Oxide (Drinklear Powder, China Chemical & Pharmaceutical Co., Ltd., Taiwan) as the bowel preparation for colonoscopy.
  Arms: Niflec

SUMMARY:
This study aims to compare the intestinal cleansing efficacy, safety, tolerability, and acceptability of sodium picosulfate/magnesium citrate and polyethylene glycol in Taiwan.

DETAILED DESCRIPTION:
Background： The quality of bowel cleansing is crucial for the quality of colonoscopy. However, the ideal bowel cleansing agent and dosage have not been determined. According to the European Society of Gastrointestinal Endoscopy (ESGE) Guideline on Bowel Preparation for Colonoscopy, published in 2013, it is recommended to use a split regimen with 4 liters of polyethylene glycol (4 L PEG) solution (or a same-day regimen for afternoon colonoscopy) for routine bowel preparation. The split regimen, especially with 2 L PEG plus ascorbate or sodium picosulfate with magnesium citrate, may be an effective alternative, especially for selective outpatient colonoscopy. For patients with renal failure, polyethylene glycol is the only recommended bowel cleansing agent.

Furthermore, patient compliance with bowel cleansing agents is of paramount importance. Drinklear powder belongs to the sodium picosulfate/magnesium citrate/magnesium oxide class of bowel cleansing agents, while Niflec Powder belongs to the polyethylene glycol class. This study aims to compare the bowel cleansing efficacy, safety, tolerability, and acceptability of sodium picosulfate/magnesium citrate/magnesium oxide and polyethylene glycol. It is a non-inferiority study conducted at a single center in Taiwan. Similar studies have been conducted both nationally and internationally, such as the study by Seo, S.I., Kang, J.G., Kim, H.S. et al. Efficacy and tolerability of 2-L polyethylene glycol with ascorbic acid versus sodium picosulfate with magnesium citrate: a randomized controlled trial. Int J Colorectal Dis 33, 541-548 (2018). https://doi.org/10.1007/s00384-018-2989-7) and The Bowklean Study in Taiwan (Hung, SY., Chen, HC. & Chen, W.TL. A Randomized Trial Comparing the Bowel Cleansing Efficacy of Sodium Picosulfate/Magnesium Citrate and Polyethylene Glycol/Bisacodyl (The Bowklean Study). Sci Rep 10, 5604 (2020). https://doi.org/10.1038/s41598-020-62120-w), which compared sodium picosulfate/magnesium citrate to polyethylene glycol/bisacodyl. Drinklear powder is similar in composition to Bowklean, but there is no direct comparative data available in Taiwan for polyethylene glycol and sodium picosulfate/magnesium citrate/magnesium oxide.

Study Design： Our hospital invites outpatient patients aged 20 to 75 years who are scheduled to undergo colonoscopy and are willing to participate in this research study. After obtaining informed consent and signing the consent form, participants will be randomly assigned to receive either Polyethylene Glycol (Niflec Powder, China Chemical & Pharmaceutical Co., Ltd., Taiwan) or Picosulfate Sodium/Citric Acid/Magnesium Oxide (Drinklear Powder, China Chemical & Pharmaceutical Co., Ltd., Taiwan) as the bowel preparation for colonoscopy. Patient data, including gender, age, medication compliance, medication acceptability, medication tolerance, safety, and bowel cleansing effectiveness, will be collected and stored at the endoscopy center. Bowel cleansing effectiveness will be assessed using the Aronchick Scale as the primary outcome, and the assessment will be performed by the gastroenterologist responsible for performing the colonoscopy of patients enrolled in the study at our hospital. Secondary outcomes will include the detection rate of colonic polyps, adenomas detection rate, safety, medication compliance, and acceptability, as well as the statistical assessment of cecal intubation success rate, cecal intubation time, and total examination time. Safety will be evaluated through the monitoring of adverse events, and tolerance and acceptability will be measured through patient questionnaires.

Methods： Subjects and Sample Size Inclusion and Exclusion Criteria for this study: Inclusion criteria include outpatient patients at our institution, aged 20 to 75 years, who are scheduled to undergo colonoscopy and are willing to participate in this research study. Exclusion criteria comprise patients with allergies to bowel preparation agents, those who fail to show up on the scheduled date, patients who refuse to participate, those unable to follow preparation instructions, individuals with intestinal perforation, gastric retention, gastrointestinal obstruction, or bowel obstruction, severe renal insufficiency (CrCl below 30 mL/min), pregnant individuals, toxic megacolon, and patients with colorectal cancer.

Statistical Analysis Plan for this study: This is a non-inferiority study with a one-sided non-inferiority hypothesis. The non-inferiority margin is set at 0.1. The sample size for each group is 220, resulting in a total of 440 participants.

Anticipated Challenges and Mitigation Strategies: Patients may be influenced by their past experiences and may be reluctant to accept the results of random allocation, leading to withdrawal from the trial. Therefore, it is crucial to provide clear explanations to patients before the trial, emphasizing that this is a randomized controlled trial. Additionally, it is important to enroll an adequate number of participants to account for potential dropouts, ensuring that the statistical goals can be achieved.

Effect： It is anticipated that the tolerability and acceptability of Drinklear Powder will be superior to Niflec Powder, and the bowel cleansing efficacy will not be inferior.

ELIGIBILITY:
Inclusion Criteria:

outpatient patients at our institution, aged 20 to 75 years, who are scheduled to undergo colonoscopy and are willing to participate in this research study.

Exclusion Criteria:

patients with allergies to bowel preparation agents, those who fail to show up on the scheduled date, patients who refuse to participate, those unable to follow preparation instructions, individuals with intestinal perforation, gastric retention, gastrointestinal obstruction, or bowel obstruction, severe renal insufficiency (CrCl below 30 mL/min), pregnant individuals, toxic megacolon, and patients with colorectal cancer.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Bowel cleansing effectiveness | 1 day
  will be assessed using the Aronchick Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Jen Catholic University Hospital, New Taipei City, Taiwan, Taiwan